CLINICAL TRIAL: NCT00486889
Title: A Long-term Study to Evaluate Growth and Development Outcomes in Patients With Infantile-Onset Pompe Disease Who Are Receiving Alglucosidase Alfa
Brief Title: Growth and Development Study of Alglucosidase Alfa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLU03606; LTS12869 (Other: Sanofi); U1111-1163-0368 (Other: UTN); 2021-005552-11 (EudraCT Number)
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Results first posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-07

CONDITIONS: Pompe Disease; Glycogen Storage Disease Type II (GSD-II); Acid Maltase Deficiency Disease
Keywords: Glycogenesis 2
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alglucosidase Alfa (Experimental): Participants received alglucosidase alfa 20 milligrams per kilogram (mg/kg) body weight as intravenous infusion every 2 weeks and were followed for 10 years or up to discontinuation from study treatment due to any reason.
  Interventions: Biological: alglucosidase alfa

INTERVENTIONS:
Biological: alglucosidase alfa — Dose: 20 mg/kg every 2 weeks; Route of administration: Intravenous infusion
  Other Names: Myozyme®; Lumizyme®

SUMMARY:
Pompe disease (also known as glycogen storage disease Type II) is a rare autosomal recessive metabolic muscle disease caused by the deficiency of acid α glucosidase (GAA), an enzyme that degrades lysosomal glycogen. As opposed to the exclusively cytoplasmic accumulation of glycogen that occurs in other glycogen storage disorders, Pompe disease is characterized by organelle bound (lysosomal) and extra-lysosomal accumulation of glycogen in many body tissues, ultimately leading to multisystemic pathology. The overall objective of this study was to evaluate the long-term growth and development of participants with infantile-onset Pompe disease with alglucosidase alfa before 1 year of age. Participants were to be followed for a 10-year period.

ELIGIBILITY:
Inclusion Criteria:

* The participant or participant's legal guardian must have provided signed, informed consent prior to performing any study-related procedures.
* The participant must have had a confirmed diagnosis of Pompe disease as determined by deficient endogenous GAA activity or GAA mutation analysis.
* The participant must be less than (<) 1 year of age at time of study enrollment (and received alglucosidase alfa treatment before 1 year of age), or the participant must be between 1 year and 24 months of age and must have had initiated alglucosidase alfa treatment prior to turning 1 year of age.

Exclusion Criteria:

* The participant was participating in another clinical study using alglucosidase alfa or any investigational therapy.

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2008-08-26 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (3):
- United States (3):
  - Gainesville, Florida
  - Decatur, Georgia
  - Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 active sites in United States. A total of 12 participants were screened from 26-August-2008 to 07-February-2014.
Pre-assignment Details: All 12 participants were enrolled and treated in the study.
Period: Overall Study
Arm/Group | Alglucosidase Alfa
Started | 12
Completed | 1
Not Completed | 11
Not completed — Death | 3
Not completed — Non-compliant | 2
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: Analysis was performed on full analysis set (FAS) that included all enrolled participants who had received at least one infusion (complete or partial) of alglucosidase alfa.
Groups:
- Alglucosidase Alfa: Participants received alglucosidase alfa 20 mg/kg body weight as intravenous infusion every 2 weeks and were followed for 10 years or up to discontinuation from study treatment due to any reason.
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: months] | 11.558 (6.226)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Recumbent Height/Length of Participants at Baseline [Mean (Standard Deviation); unit: centimeter (cm)] | 72.95 (10.24)
Body Weight of Participants at Baseline [Mean (Standard Deviation); unit: kilogram (Kg)] | 8.42 (2.61)
Head Circumference of Participants at Baseline [Mean (Standard Deviation); unit: cm] | 45.20 (3.61)

OUTCOME MEASURES:

1. Primary Outcome: Recumbent Height/Length of Participants in Centimeters (cm)
Description: Height/Length of Participants was measured in centimeters. Week is denoted as Wk in time frame section.
Time Frame: Participants 1-12:Baseline, Participant1: Wk 52, Participant2: Wk82, Participants 3-4: Wk208, Participant5: Wk12, Participant6: Wk365, Participant7: Wk64, Participant8:Wk156, Participant9:Wk364, Participant10:Wk52, Participant11:Wk156, Participant12:Wk520
Population: Analysis was performed on FAS population. No summary analysis was done and participant wise data were reported at available specified timepoints.
Measure: Number; unit: cm
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 12
cm
  Participant-1 Baseline: number analyzed (Participants) | 1
  Participant-1 Baseline | 80.4
  Participant-1 Week 52: number analyzed (Participants) | 1
  Participant-1 Week 52 | 93.8
  Participant-2 Baseline: number analyzed (Participants) | 1
  Participant-2 Baseline | 67.7
  Participant-2 Week 82: number analyzed (Participants) | 1
  Participant-2 Week 82 | 91.1
  Participant-3 Baseline: number analyzed (Participants) | 1
  Participant-3 Baseline | 69.1
  Participant-3 Week 208: number analyzed (Participants) | 1
  Participant-3 Week 208 | 107.5
  Participant-4 Baseline: number analyzed (Participants) | 1
  Participant-4 Baseline | 67.0
  Participant-4 Week 208: number analyzed (Participants) | 1
  Participant-4 Week 208 | 110.0
  Participant-5 Baseline: number analyzed (Participants) | 1
  Participant-5 Baseline | 71.4
  Participant-5 Week 12: number analyzed (Participants) | 1
  Participant-5 Week 12 | 71.1
  Participant-6 Baseline: number analyzed (Participants) | 1
  Participant-6 Baseline | 83.5
  Participant-6 Week 365: number analyzed (Participants) | 1
  Participant-6 Week 365 | 131.0
  Participant-7 Baseline: number analyzed (Participants) | 1
  Participant-7 Baseline | 57.2
  Participant-7 Week 64: number analyzed (Participants) | 1
  Participant-7 Week 64 | 80.5
  Participant-8 Baseline: number analyzed (Participants) | 1
  Participant-8 Baseline | 70.4
  Participant-8 Week 156: number analyzed (Participants) | 1
  Participant-8 Week 156 | 110.3
  Participant-9 Baseline: number analyzed (Participants) | 1
  Participant-9 Baseline | 61.0
  Participant-9 Week 364: number analyzed (Participants) | 1
  Participant-9 Week 364 | 117.0
  Participant-10 Baseline: number analyzed (Participants) | 1
  Participant-10 Baseline | 76.7
  Participant-10 Week 52: number analyzed (Participants) | 1
  Participant-10 Week 52 | 83.8
  Participant-11 Baseline: number analyzed (Participants) | 1
  Participant-11 Baseline | 95.0
  Participant-11 Week 156: number analyzed (Participants) | 1
  Participant-11 Week 156 | 115.0
  Participant-12 Baseline: number analyzed (Participants) | 1
  Participant-12 Baseline | 76.0
  Participant-12 Week 520: number analyzed (Participants) | 1
  Participant-12 Week 520 | 139.7

2. Primary Outcome: Body Weight of Participants in Kilograms (kg)
Description: Body Weight of Participants was measured in Kilograms (kg). Week is denoted as Wk in time frame section.
Time Frame: Participant1-12:Baseline, Participant1:Wk 52, Participant2:Wk82, Participant3: Wk208,Participant4:Wk364,Participant5:Wk12,Participant6:Wk365,Participant7:Wk64,Participant8:Wk156,Participant9:Wk364,Participant10:Wk52,Participant11:Wk156,Participant12:Wk520
Population: as for outcome 1
Measure: Number; unit: kilograms
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 12
kilograms
  Participant-1 Baseline: number analyzed (Participants) | 1
  Participant-1 Baseline | 10.0
  Participant-1 Week 52: number analyzed (Participants) | 1
  Participant-1 Week 52 | 13.8
  Participant-2 Baseline: number analyzed (Participants) | 1
  Participant-2 Baseline | 8.0
  Participant-2 Week 82: number analyzed (Participants) | 1
  Participant-2 Week 82 | 13.1
  Participant-3 Baseline: number analyzed (Participants) | 1
  Participant-3 Baseline | 6.5
  Participant-3 Week 208: number analyzed (Participants) | 1
  Participant-3 Week 208 | 17.4
  Participant-4 Baseline: number analyzed (Participants) | 1
  Participant-4 Baseline | 6.2
  Participant-4 Week 364: number analyzed (Participants) | 1
  Participant-4 Week 364 | 33.3
  Participant-5 Baseline: number analyzed (Participants) | 1
  Participant-5 Baseline | 6.5
  Participant-5 Week 12: number analyzed (Participants) | 1
  Participant-5 Week 12 | 6.7
  Participant-6 Baseline: number analyzed (Participants) | 1
  Participant-6 Baseline | 12.8
  Participant-6 Week 365: number analyzed (Participants) | 1
  Participant-6 Week 365 | 47.5
  Participant-7 Baseline: number analyzed (Participants) | 1
  Participant-7 Baseline | 5.0
  Participant-7 Week 64: number analyzed (Participants) | 1
  Participant-7 Week 64 | 12.2
  Participant-8 Baseline: number analyzed (Participants) | 1
  Participant-8 Baseline | 8.9
  Participant-8 Week 156: number analyzed (Participants) | 1
  Participant-8 Week 156 | 20.3
  Participant-9 Baseline: number analyzed (Participants) | 1
  Participant-9 Baseline | 5.2
  Participant-9 Week 364: number analyzed (Participants) | 1
  Participant-9 Week 364 | 23.1
  Participant-10 Baseline: number analyzed (Participants) | 1
  Participant-10 Baseline | 10.5
  Participant-10 Week 52: number analyzed (Participants) | 1
  Participant-10 Week 52 | 12.8
  Participant-11 Baseline: number analyzed (Participants) | 1
  Participant-11 Baseline | 12.1
  Participant-11 Week 156: number analyzed (Participants) | 1
  Participant-11 Week 156 | 35.0
  Participant-12 Baseline: number analyzed (Participants) | 1
  Participant-12 Baseline | 9.3
  Participant-12 Week 520: number analyzed (Participants) | 1
  Participant-12 Week 520 | 46.3

3. Primary Outcome: Head Circumference of Participants in Centimeters (cm)
Description: Head Circumference of Participants was measured in Centimeters.
Time Frame: Participants1-12:Baseline, Participant1:Week(Wk)52, Participant2:Wk82, Participants3and4:Wk208, Participant5:Wk12, Participant6:Wk365, Participant7:Wk64, Participant8:Wk156, Participant9:Wk312, Participant10:Wk52, Participant11:Wk156, Participant12:Wk468
Population: as for outcome 1
Measure: Number; unit: cm
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 12
cm
  Participant-1 Baseline: number analyzed (Participants) | 1
  Participant-1 Baseline | 45.3
  Participant-1 Week 52: number analyzed (Participants) | 1
  Participant-1 Week 52 | 48.1
  Participant-2 Baseline: number analyzed (Participants) | 1
  Participant-2 Baseline | 44.0
  Participant-2 Week 82: number analyzed (Participants) | 1
  Participant-2 Week 82 | 49.3
  Participant-3 Baseline: number analyzed (Participants) | 1
  Participant-3 Baseline | 43.4
  Participant-3 Week 208: number analyzed (Participants) | 1
  Participant-3 Week 208 | 52.8
  Participant-4 Baseline: number analyzed (Participants) | 1
  Participant-4 Baseline | 42.6
  Participant-4 Week 208: number analyzed (Participants) | 1
  Participant-4 Week 208 | 52.4
  Participant-5 Baseline: number analyzed (Participants) | 1
  Participant-5 Baseline | 44.3
  Participant-5 Week 12: number analyzed (Participants) | 1
  Participant-5 Week 12 | 44.5
  Participant-6 Baseline: number analyzed (Participants) | 1
  Participant-6 Baseline | 49.9
  Participant-6 Week 365: number analyzed (Participants) | 1
  Participant-6 Week 365 | 56.3
  Participant-7 Baseline: number analyzed (Participants) | 1
  Participant-7 Baseline | 39.6
  Participant-7 Week 64: number analyzed (Participants) | 1
  Participant-7 Week 64 | 48.0
  Participant-8 Baseline: number analyzed (Participants) | 1
  Participant-8 Baseline | 50.8
  Participant-8 Week 156: number analyzed (Participants) | 1
  Participant-8 Week 156 | 54.0
  Participant-9 Baseline: number analyzed (Participants) | 1
  Participant-9 Baseline | 40.0
  Participant-9 Week 312: number analyzed (Participants) | 1
  Participant-9 Week 312 | 52.0
  Participant-10 Baseline: number analyzed (Participants) | 1
  Participant-10 Baseline | 48.5
  Participant-10 Week 52: number analyzed (Participants) | 1
  Participant-10 Week 52 | 49.5
  Participant-11 Baseline: number analyzed (Participants) | 1
  Participant-11 Baseline | 48.0
  Participant-11 Week 156: number analyzed (Participants) | 1
  Participant-11 Week 156 | 50.8
  Participant-12 Baseline: number analyzed (Participants) | 1
  Participant-12 Baseline | 46.0
  Participant-12 Week 468: number analyzed (Participants) | 1
  Participant-12 Week 468 | 56.0

4. Primary Outcome: Motor Subscale of Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) Normative Composite Scores
Description: Bayley-III: Instrument designed to measure developmental functioning of infants and toddlers between ages of 1 and 42 months (age adjustments for prematurity are accommodated with tool). Bayley-III administered up to 42 months of age and provides age specific norm-referenced composite scores for cognitive scales (91 items, composite score minimum 55 and maximum 145), language scale (98 items, composite score minimum 47 and maximum 153), motor scale (138 items, composite score minimum 46 and maximum 154) skills. For all raw scores (for scales), higher scores indicates greater number of developmental skills credited. For norm-based composite scales for motor scale, score of 100 defines average performance of given age group, scores of 85 and 115 are 1 standard deviation (SD) below an above mean, respectively, and scores of 70 and 130 are equivalent to 2 SD from mean.
Time Frame: Participants 1-12: Baseline, Participant-1: Week 52, Participant-2: Week 83, Participants 3 and 4: Week 104, Participant-6: Week 78, Participants 7 and 8: Week 26, Participant-9: Week 156, Participants 10 and 11: Week 26, Participant-12: Week 104
Population: as for outcome 1
Measure: Number; unit: score on a scale
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 12
score on a scale
  Participant-1 Baseline: number analyzed (Participants) | 1
  Participant-1 Baseline | 94
  Participant-1 Week 52: number analyzed (Participants) | 1
  Participant-1 Week 52 | 94
  Participant-2 Baseline: number analyzed (Participants) | 1
  Participant-2 Baseline | 94
  Participant-2 Week 83: number analyzed (Participants) | 1
  Participant-2 Week 83 | 91
  Participant-3 Baseline: number analyzed (Participants) | 1
  Participant-3 Baseline | 46
  Participant-3 Week 104: number analyzed (Participants) | 1
  Participant-3 Week 104 | 46
  Participant-4 Baseline: number analyzed (Participants) | 1
  Participant-4 Baseline | 46
  Participant-4 Week 104: number analyzed (Participants) | 1
  Participant-4 Week 104 | 46
  Participant-5 Baseline: number analyzed (Participants) | 1
  Participant-5 Baseline | 58
  Participant-6 Baseline: number analyzed (Participants) | 1
  Participant-6 Baseline | 79
  Participant-6 Week 78: number analyzed (Participants) | 1
  Participant-6 Week 78 | 100
  Participant-7 Baseline: number analyzed (Participants) | 1
  Participant-7 Baseline | 61
  Participant-7 Week 26: number analyzed (Participants) | 1
  Participant-7 Week 26 | 46
  Participant-8 Baseline: number analyzed (Participants) | 1
  Participant-8 Baseline | 46
  Participant-8 Week 26: number analyzed (Participants) | 1
  Participant-8 Week 26 | 46
  Participant-9 Baseline: number analyzed (Participants) | 1
  Participant-9 Baseline | 46
  Participant-9 Week 156: number analyzed (Participants) | 1
  Participant-9 Week 156 | 70
  Participant-10 Baseline: number analyzed (Participants) | 1
  Participant-10 Baseline | 61
  Participant-10 Week 26: number analyzed (Participants) | 1
  Participant-10 Week 26 | 73
  Participant-11 Baseline: number analyzed (Participants) | 1
  Participant-11 Baseline | 61
  Participant-11 Week 26: number analyzed (Participants) | 1
  Participant-11 Week 26 | 58
  Participant-12 Baseline: number analyzed (Participants) | 1
  Participant-12 Baseline | 55
  Participant-12 Week 104: number analyzed (Participants) | 1
  Participant-12 Week 104 | 61

5. Primary Outcome: Gross Motor Function Measure (GMFM-88) Total Scores
Description: GMFM-88 is developed specifically to detect quantitative changes in gross motor function that consists of 88 items organized into 5 dimensions: lying and rolling, sitting, crawling and kneeling, standing, and walking, running and jumping. Each item is scored on a 4-point Likert scale that ranges from 0 to 3, i.e., 0=cannot do; 1=initiated (less than [<] 10 percent [%] of task); 2=partially completed (10 to <100% of task); 3=task completion. The score for each dimension is expressed as percentage of the maximum score for that dimension. Total GMFM-88 score is obtained by adding percentage score for each dimension and dividing the sum by total number of dimensions. Total score ranges from 0 to 100, where higher score indicates better gross motor functions.
Time Frame: Participants 1-12: Baseline, Participants 1 and 2: Wk 52, Participants 3 and 4: Wk 208, Participant-6: Wk 359, Participant-7: Wk 26, Participant-8: Wk 156, Participant-9: Wk 312, Participant-11: Wk 156, Participant-12: Wk416
Population: as for outcome 1
Measure: Number; unit: score on a scale
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 12
score on a scale
  Participant-1 Baseline: number analyzed (Participants) | 1
  Participant-1 Baseline | 27.98
  Participant-1 Week 52: number analyzed (Participants) | 1
  Participant-1 Week 52 | 59.65
  Participant-2 Baseline: number analyzed (Participants) | 1
  Participant-2 Baseline | 32.42
  Participant-2 Week 52: number analyzed (Participants) | 1
  Participant-2 Week 52 | 91.52
  Participant-3 Baseline: number analyzed (Participants) | 1
  Participant-3 Baseline | 7.16
  Participant-3 Week 208: number analyzed (Participants) | 1
  Participant-3 Week 208 | 2.75
  Participant-4 Baseline: number analyzed (Participants) | 1
  Participant-4 Baseline | 2.18
  Participant-4 Week 208: number analyzed (Participants) | 1
  Participant-4 Week 208 | 0.39
  Participant-5 Baseline: number analyzed (Participants) | 1
  Participant-5 Baseline | 12.39
  Participant-6 Baseline: number analyzed (Participants) | 1
  Participant-6 Baseline | 62.22
  Participant-6 Week 359: number analyzed (Participants) | 1
  Participant-6 Week 359 | 97.11
  Participant-7 Baseline: number analyzed (Participants) | 1
  Participant-7 Baseline | 8.27
  Participant-7 Week 26: number analyzed (Participants) | 1
  Participant-7 Week 26 | 15.83
  Participant-8 Baseline: number analyzed (Participants) | 1
  Participant-8 Baseline | 0.39
  Participant-8 Week 156: number analyzed (Participants) | 1
  Participant-8 Week 156 | 0.39
  Participant-9 Baseline: number analyzed (Participants) | 1
  Participant-9 Baseline | 2.35
  Participant-9 Week 312: number analyzed (Participants) | 1
  Participant-9 Week 312 | 88.23
  Participant-10 Baseline: number analyzed (Participants) | 1
  Participant-10 Baseline | 34.43
  Participant-11 Baseline: number analyzed (Participants) | 1
  Participant-11 Baseline | 16.71
  Participant-11 Week 156: number analyzed (Participants) | 1
  Participant-11 Week 156 | 9.86
  Participant-12 Baseline: number analyzed (Participants) | 1
  Participant-12 Baseline | 21.94
  Participant-12 Week 416: number analyzed (Participants) | 1
  Participant-12 Week 416 | 27.39

6. Primary Outcome: Pompe Pediatric Evaluation of Disability Inventory (Pompe PEDI) Scaled Scores
Description: Pompe PEDI is disease specific version of PEDI developed to assess functional capabilities and performance in children with Pompe disease from 2 months up to adolescence. It consists of all items of original PEDI Functional Skills Scales and Caregiver Assistance Scales for three content domains: self-care, mobility, and social function. Additional items were added to Functional Skills Scales Mobility and Self-care domains. Norm-based scoring is developed for additional items and scoring algorithms for PEDI are adjusted to reflect normative data collected for Pompe PEDI. Scaled scores for each domain range from 0-100 and provide indication of performance of child along continuum of relatively easy to relatively difficult items in particular domain of PEDI, where higher score indicates increased degrees of functional performance.
Time Frame: Participants1-12:Baseline, Participants 1 and 2: Wk 52, Participants 3 and 4: Wk 208, Participant-6: Wk 359, Participant-7: Wk 52, Participant-8: Wk156, Participant-9: Wk 312, Participant-10: Wk 26, Participant-11: Wk 156, Participant-12: Wk 416
Population: Analysis was preformed on FAS population. No summary analysis was done and participant wise data were reported at available specified timepoint.
Measure: Number; unit: score on a scale
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 12
score on a scale
  Participant-1 Baseline: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-1 Baseline: Functional Skills- Self-Care | 40.62
  Participant-1 Week 52: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-1 Week 52: Functional Skills- Self-Care | 50.15
  Participant-1 Baseline: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-1 Baseline: Caregiver Assistance- Self-Care | 0
  Participant-1 Week 52: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-1 Week 52: Caregiver Assistance- Self-Care | 20.1
  Participant-1 Baseline: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-1 Baseline: Functional Skills- Mobility | 39.68
  Participant-1 Week 52: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-1 Week 52: Functional Skills- Mobility | 56.31
  Participant-1 Baseline: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-1 Baseline: Caregiver Assistance- Mobility | 42.7
  Participant-1 Week 52: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-1 Week 52: Caregiver Assistance- Mobility | 47.2
  Participant-1 Baseline: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-1 Baseline: Functional Skills- Social | 36.1
  Participant-1 Week 52: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-1 Week 52: Functional Skills- Social | 45
  Participant-1 Baseline: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-1 Baseline: Caregiver Assistance- Social | 35.9
  Participant-1 Week 52: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-1 Week 52: Caregiver Assistance- Social | 31.6
  Participant-2 Baseline: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-2 Baseline: Functional Skills- Self-Care | 23.05
  Participant-2 Week 52: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-2 Week 52: Functional Skills- Self-Care | 59.79
  Participant-2 Week 52: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-2 Week 52: Caregiver Assistance- Self-Care | 32.3
  Participant-2 Baseline: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-2 Baseline: Functional Skills- Mobility | 28.81
  Participant-2 Week 52: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-2 Week 52: Functional Skills- Mobility | 62.11
  Participant-2 Week 52: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-2 Week 52: Caregiver Assistance- Mobility | 72.7
  Participant-2 Week 52: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-2 Week 52: Functional Skills- Social | 52
  Participant-3 Baseline: Functional Skills-Self-Care: number analyzed (Participants) | 1
  Participant-3 Baseline: Functional Skills-Self-Care | 21.03
  Participant-3 Week 208: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-3 Week 208: Functional Skills- Self-Care | 34.24
  Participant-3 Baseline: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-3 Baseline: Caregiver Assistance- Self-Care | 11.6
  Participant-3 Week 208: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-3 Week 208: Caregiver Assistance- Self-Care | 0
  Participant-3 Baseline: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-3 Baseline: Functional Skills- Mobility | 15.06
  Participant-3 Week 208: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-3 Week 208: Functional Skills- Mobility | 4.53
  Participant-3 Baseline: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-3 Baseline: Caregiver Assistance- Mobility | 0
  Participant-3 Week 208: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-3 Week 208: Caregiver Assistance- Mobility | 0
  Participant-3 Baseline: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-3 Baseline: Functional Skills- Social | 21.6
  Participant-3 Week 208: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-3 Week 208: Functional Skills- Social | 40.4
  Participant-3 Baseline: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-3 Baseline: Caregiver Assistance- Social | 0
  Participant-3 Week 208: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-3 Week 208: Caregiver Assistance- Social | 11.3
  Participant-4 Baseline: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-4 Baseline: Functional Skills- Self-Care | 4.92
  Participant-4 Week 208: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-4 Week 208: Functional Skills- Self-Care | 23.05
  Participant-4 Baseline: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-4 Baseline: Caregiver Assistance- Self-Care | 0
  Participant-4 Week 208: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-4 Week 208: Caregiver Assistance- Self-Care | 0
  Participant-4 Baseline: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-4 Baseline: Functional Skills- Mobility | 4.53
  Participant-4 Week 208: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-4 Week 208: Functional Skills- Mobility | 0
  Participant-4 Baseline: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-4 Baseline: Caregiver Assistance- Mobility | 0
  Participant-4 Week 208: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-4 Week 208: Caregiver Assistance- Mobility | 0
  Participant-4 Baseline: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-4 Baseline: Functional Skills- Social | 14.7
  Participant-4 Week 208: Functional Skills-Social: number analyzed (Participants) | 1
  Participant-4 Week 208: Functional Skills-Social | 40.4
  Participant-4 Baseline: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-4 Baseline: Caregiver Assistance- Social | 0
  Participant-4 Week 208: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-4 Week 208: Caregiver Assistance- Social | 11.3
  Participant-5 Baseline: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-5 Baseline: Functional Skills- Self-Care | 36.16
  Participant-5 Baseline: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-5 Baseline: Caregiver Assistance- Self-Care | 0
  Participant-5 Baseline: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-5 Baseline: Functional Skills- Mobility | 19.75
  Participant-5 Baseline: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-5 Baseline: Caregiver Assistance- Mobility | 0
  Participant-5 Baseline: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-5 Baseline: Functional Skills- Social | 32.9
  Participant-5 Baseline: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-5 Baseline: Caregiver Assistance- Social | 0
  Participant-6 Baseline: Functional Skills-Self-Care: number analyzed (Participants) | 1
  Participant-6 Baseline: Functional Skills-Self-Care | 45.7
  Participant-6 Week 359: Functional Skills-Self-Care: number analyzed (Participants) | 1
  Participant-6 Week 359: Functional Skills-Self-Care | 81.36
  Participant-6 Baseline: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-6 Baseline: Caregiver Assistance- Self-Care | 44.4
  Participant-6 Week 359: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-6 Week 359: Caregiver Assistance- Self-Care | 100
  Participant-6 Baseline: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-6 Baseline: Functional Skills- Mobility | 52.44
  Participant-6 Week 359: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-6 Week 359: Functional Skills- Mobility | 76.46
  Participant-6 Baseline: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-6 Baseline: Caregiver Assistance- Mobility | 61.8
  Participant-6 Week 359: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-6 Week 359: Caregiver Assistance- Mobility | 100
  Participant-6 Baseline: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-6 Baseline: Functional Skills- Social | 40.4
  Participant-6 Week 359: Functional Skills-Social: number analyzed (Participants) | 1
  Participant-6 Week 359: Functional Skills-Social | 100
  Participant-6 Baseline: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-6 Baseline: Caregiver Assistance- Social | 57.3
  Participant-6 Week 359: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-6 Week 359: Caregiver Assistance- Social | 100
  Participant-7 Baseline: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-7 Baseline: Functional Skills- Self-Care | 12.7
  Participant-7 Week 52: Functional Skills-Self-Care: number analyzed (Participants) | 1
  Participant-7 Week 52: Functional Skills-Self-Care | 33.1
  Participant-7 Week 52: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-7 Week 52: Caregiver Assistance- Self-Care | 11.6
  Participant-7 Baseline: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-7 Baseline: Functional Skills- Mobility | 4.53
  Participant-7 Week 52: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-7 Week 52: Functional Skills- Mobility | 25.12
  Participant-7 Baseline: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-7 Baseline: Caregiver Assistance- Mobility | 0
  Participant-7 Week 52: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-7 Week 52: Caregiver Assistance- Mobility | 0
  Participant-7 Baseline: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-7 Baseline: Functional Skills- Social | 6.6
  Participant-7 Week 52: Functional Skills-Social: number analyzed (Participants) | 1
  Participant-7 Week 52: Functional Skills-Social | 27.7
  Participant-7 Baseline: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-7 Baseline: Caregiver Assistance- Social | 0
  Participant-7 Week 52: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-7 Week 52: Caregiver Assistance- Social | 0
  Participant-8 Baseline: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-8 Baseline: Functional Skills- Self-Care | 0.01
  Participant-8 Week 156: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-8 Week 156: Functional Skills- Self-Care | 12.7
  Participant-8 Baseline: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-8 Baseline: Caregiver Assistance- Self-Care | 0
  Participant-8 Week 156: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-8 Week 156: Caregiver Assistance- Self-Care | 0
  Participant-8 Baseline: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-8 Baseline: Functional Skills- Mobility | 0.01
  Participant-8 Week 156: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-8 Week 156: Functional Skills- Mobility | 0
  Participant-8 Baseline: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-8 Baseline: Caregiver Assistance- Mobility | 0
  Participant-8 Week 156: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-8 Week 156: Caregiver Assistance- Mobility | 0
  Participant-8 Baseline: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-8 Baseline: Functional Skills- Social | 3.1
  Participant-8 Week 156: Functional Skills-Social: number analyzed (Participants) | 1
  Participant-8 Week 156: Functional Skills-Social | 35.1
  Participant-8 Baseline: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-8 Baseline: Caregiver Assistance- Social | 0
  Participant-8 Week 156: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-8 Week 156: Caregiver Assistance- Social | 20.4
  Participant-9 Baseline: Functional Skills-Self-Care: number analyzed (Participants) | 1
  Participant-9 Baseline: Functional Skills-Self-Care | 16.09
  Participant-9 Week 312: Functional Skills-Self-Care: number analyzed (Participants) | 1
  Participant-9 Week 312: Functional Skills-Self-Care | 77.1
  Participant-9 Baseline: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-9 Baseline: Caregiver Assistance- Self-Care | 0
  Participant-9 Week 312: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-9 Week 312: Caregiver Assistance- Self-Care | 100
  Participant-9 Baseline: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-9 Baseline: Functional Skills- Mobility | 4.53
  Participant-9 Week 312: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-9 Week 312: Functional Skills- Mobility | 63.25
  Participant-9 Baseline: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-9 Baseline: Caregiver Assistance- Mobility | 0
  Participant-9 Week 312 :Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-9 Week 312 :Caregiver Assistance- Mobility | 100
  Participant-9 Baseline: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-9 Baseline: Functional Skills- Social | 10.5
  Participant-9 Week 312: Functional Skills-Social: number analyzed (Participants) | 1
  Participant-9 Week 312: Functional Skills-Social | 73.4
  Participant-9 Baseline: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-9 Baseline: Caregiver Assistance- Social | 0
  Participant-9 Week 312: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-9 Week 312: Caregiver Assistance- Social | 100
  Participant-10 Baseline: Functional Skills-Self-Care: number analyzed (Participants) | 1
  Participant-10 Baseline: Functional Skills-Self-Care | 35.25
  Participant-10 Week 26: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-10 Week 26: Functional Skills- Self-Care | 49.18
  Participant-10 Baseline: Caregiver Assistance Self-Care: number analyzed (Participants) | 1
  Participant-10 Baseline: Caregiver Assistance Self-Care | 11.6
  Participant-10 Week 26: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-10 Week 26: Caregiver Assistance- Self-Care | 42.8
  Participant-10 Baseline: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-10 Baseline: Functional Skills- Mobility | 34.55
  Participant-10 Week 26: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-10 Week 26: Functional Skills- Mobility | 49.26
  Participant-10 Baseline: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-10 Baseline: Caregiver Assistance- Mobility | 31.9
  Participant-10 Week 26: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-10 Week 26: Caregiver Assistance- Mobility | 48.5
  Participant-10 Baseline: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-10 Baseline: Functional Skills- Social | 31.6
  Participant-10 Week 26: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-10 Week 26: Functional Skills- Social | 44.4
  Participant-10 Baseline: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-10 Baseline: Caregiver Assistance- Social | 11.3
  Participant-10 Week 26: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-10 Week 26: Caregiver Assistance- Social | 50.9
  Participant-11 Baseline: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-11 Baseline: Functional Skills- Self-Care | 43.58
  Participant-11 Week 156: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-11 Week 156: Functional Skills- Self-Care | 43
  Participant-11 Baseline: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-11 Baseline: Caregiver Assistance- Self-Care | 25.4
  Participant-11 Week 156: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-11 Week 156: Caregiver Assistance- Self-Care | 25.4
  Participant-11 Baseline: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-11 Baseline: Functional Skills- Mobility | 28.15
  Participant-11 Week 156: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-11 Week 156: Functional Skills- Mobility | 25.93
  Participant-11 Baseline: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-11 Baseline: Caregiver Assistance- Mobility | 0
  Participant-11 Week 156: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-11 Week 156: Caregiver Assistance- Mobility | 11.7
  Participant-11 Baseline: Functional Skills-Social: number analyzed (Participants) | 1
  Participant-11 Baseline: Functional Skills-Social | 37
  Participant-11 Week 156: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-11 Week 156: Functional Skills- Social | 51.4
  Participant-11 Baseline: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-11 Baseline: Caregiver Assistance- Social | 11.3
  Participant-11 Week 156: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-11 Week 156: Caregiver Assistance- Social | 39.6
  Participant-12 Baseline: Functional Skills- Self-Care: number analyzed (Participants) | 1
  Participant-12 Baseline: Functional Skills- Self-Care | 31.8
  Participant-12 Week 416: Functional Skills-Self-Care: number analyzed (Participants) | 1
  Participant-12 Week 416: Functional Skills-Self-Care | 64.08
  Participant-12 Baseline: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-12 Baseline: Caregiver Assistance- Self-Care | 11.6
  Participant-12 Week 416: Caregiver Assistance- Self-Care: number analyzed (Participants) | 1
  Participant-12 Week 416: Caregiver Assistance- Self-Care | 55.7
  Participant-12 Baseline: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-12 Baseline: Functional Skills- Mobility | 26.71
  Participant-12 Week 416: Functional Skills- Mobility: number analyzed (Participants) | 1
  Participant-12 Week 416: Functional Skills- Mobility | 48.06
  Participant-12 Baseline: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-12 Baseline: Caregiver Assistance- Mobility | 11.7
  Participant-12 Week 416: Caregiver Assistance- Mobility: number analyzed (Participants) | 1
  Participant-12 Week 416: Caregiver Assistance- Mobility | 40.9
  Participant-12 Baseline: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-12 Baseline: Functional Skills- Social | 37.9
  Participant-12 Week 416: Functional Skills- Social: number analyzed (Participants) | 1
  Participant-12 Week 416: Functional Skills- Social | 73.4
  Participant-12 Baseline: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-12 Baseline: Caregiver Assistance- Social | 11.3
  Participant-12 Week 416: Caregiver Assistance- Social: number analyzed (Participants) | 1
  Participant-12 Week 416: Caregiver Assistance- Social | 63.3

7. Primary Outcome: Cognitive and Language Subscales of Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) Normative Composite Scores
Description: Bayley-III: Instrument designed to measure developmental functioning of infants and toddlers between ages of 1 and 42 months (age adjustments for prematurity are accommodated with tool). Bayley-III administered up to 42 months of age and provides age specific norm-referenced composite scores for cognitive scales (91 items, composite score minimum 55 and maximum 145), language scale (98 items, composite score minimum 47 and maximum 153), motor scale (138 items, composite score minimum 46 and maximum 154) skills. For all raw scores (for scales), higher scores indicates greater number of developmental skills credited. For norm-based composite scales for cognitive and language, score of 100 defines average performance of given age group, scores of 85 and 115 are 1 SD below an above mean, respectively, and scores of 70 and 130 are equivalent to 2 SD from mean.
Time Frame: Participants 1-12: Baseline, Participant-1: Week 52, Participant-2: Week 83, Participants 3 and 4: Week 104, Participant-6: Week 78, Participants 7 and 8: Week 26, Participant-9: Week 156, Participants 10 and 11:Week 26, Participant-12: Week 104
Population: as for outcome 1
Measure: Number; unit: score on a scale
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 12
score on a scale
  Participant-1 Baseline: Cognitive: number analyzed (Participants) | 1
  Participant-1 Baseline: Cognitive | 90
  Participant-1 Week 52: Cognitive: number analyzed (Participants) | 1
  Participant-1 Week 52: Cognitive | 100
  Participant-2 Baseline: Cognitive: number analyzed (Participants) | 1
  Participant-2 Baseline: Cognitive | 85
  Participant-2 Week 83: Cognitive: number analyzed (Participants) | 1
  Participant-2 Week 83: Cognitive | 100
  Participant-3 Baseline: Cognitive: number analyzed (Participants) | 1
  Participant-3 Baseline: Cognitive | 65
  Participant-3 Week 104: Cognitive: number analyzed (Participants) | 1
  Participant-3 Week 104: Cognitive | 55
  Participant-4 Baseline: Cognitive: number analyzed (Participants) | 1
  Participant-4 Baseline: Cognitive | 55
  Participant-4 Week 104: Cognitive: number analyzed (Participants) | 1
  Participant-4 Week 104: Cognitive | 55
  Participant-5 Baseline: Cognitive: number analyzed (Participants) | 1
  Participant-5 Baseline: Cognitive | 60
  Participant-6 Baseline: Cognitive: number analyzed (Participants) | 1
  Participant-6 Baseline: Cognitive | 75
  Participant-6 Week 78: Cognitive: number analyzed (Participants) | 1
  Participant-6 Week 78: Cognitive | 105
  Participant-7 Baseline: Cognitive: number analyzed (Participants) | 1
  Participant-7 Baseline: Cognitive | 65
  Participant-7 Week 26: Cognitive: number analyzed (Participants) | 1
  Participant-7 Week 26: Cognitive | 60
  Participant-8 Baseline: Cognitive: number analyzed (Participants) | 1
  Participant-8 Baseline: Cognitive | 55
  Participant-8 Week 26: Cognitive: number analyzed (Participants) | 1
  Participant-8 Week 26: Cognitive | 55
  Participant-9 Baseline: Cognitive: number analyzed (Participants) | 1
  Participant-9 Baseline: Cognitive | 55
  Participant-9 Week 156: Cognitive: number analyzed (Participants) | 1
  Participant-9 Week 156: Cognitive | 65
  Participant-10 Baseline: Cognitive: number analyzed (Participants) | 1
  Participant-10 Baseline: Cognitive | 85
  Participant-10 Week 26: Cognitive: number analyzed (Participants) | 1
  Participant-10 Week 26: Cognitive | 85
  Participant-11 Baseline: Cognitive: number analyzed (Participants) | 1
  Participant-11 Baseline: Cognitive | 75
  Participant-11 Week 26: Cognitive: number analyzed (Participants) | 1
  Participant-11 Week 26: Cognitive | 75
  Participant-12 Baseline: Cognitive: number analyzed (Participants) | 1
  Participant-12 Baseline: Cognitive | 80
  Participant-12 Week 104: Cognitive: number analyzed (Participants) | 1
  Participant-12 Week 104: Cognitive | 85
  Participant-1 Baseline: Language: number analyzed (Participants) | 1
  Participant-1 Baseline: Language | 103
  Participant-1 Week 52: Language: number analyzed (Participants) | 1
  Participant-1 Week 52: Language | 103
  Participant-2 Baseline: Language: number analyzed (Participants) | 1
  Participant-2 Baseline: Language | 79
  Participant-2 Week 83: Language: number analyzed (Participants) | 1
  Participant-2 Week 83: Language | 103
  Participant-3 Baseline: Language: number analyzed (Participants) | 1
  Participant-3 Baseline: Language | 59
  Participant-3 Week 104: Language: number analyzed (Participants) | 1
  Participant-3 Week 104: Language | 53
  Participant-4 Baseline: Language: number analyzed (Participants) | 1
  Participant-4 Baseline: Language | 47
  Participant-4 Week 104: Language: number analyzed (Participants) | 1
  Participant-4 Week 104: Language | 47
  Participant-5 Baseline: Language: number analyzed (Participants) | 1
  Participant-5 Baseline: Language | 71
  Participant-6 Baseline: Language: number analyzed (Participants) | 1
  Participant-6 Baseline: Language | 71
  Participant-6 Week 78: Language: number analyzed (Participants) | 1
  Participant-6 Week 78: Language | 91
  Participant-7 Baseline: Language: number analyzed (Participants) | 1
  Participant-7 Baseline: Language | 65
  Participant-7 Week 26: Language: number analyzed (Participants) | 1
  Participant-7 Week 26: Language | 50
  Participant-8 Baseline: Language: number analyzed (Participants) | 1
  Participant-8 Baseline: Language | 47
  Participant-8 Week 26: Language: number analyzed (Participants) | 1
  Participant-8 Week 26: Language | 47
  Participant-9 Baseline: Language: number analyzed (Participants) | 1
  Participant-9 Baseline: Language | 53
  Participant-9 Week 156: Language: number analyzed (Participants) | 1
  Participant-9 Week 156: Language | 74
  Participant-10 Baseline: Language: number analyzed (Participants) | 1
  Participant-10 Baseline: Language | 94
  Participant-10 Week 26: Language: number analyzed (Participants) | 1
  Participant-10 Week 26: Language | 86
  Participant-11 Baseline: Language: number analyzed (Participants) | 1
  Participant-11 Baseline: Language | 68
  Participant-11 Week 26: Language: number analyzed (Participants) | 1
  Participant-11 Week 26: Language | 71
  Participant-12 Baseline: Language: number analyzed (Participants) | 1
  Participant-12 Baseline: Language | 86
  Participant-12 Week 104: Language: number analyzed (Participants) | 1
  Participant-12 Week 104: Language | 65

8. Primary Outcome: Brief Intelligence Quotient (IQ) Score of the Leiter International Performance Scale-Revised (Leiter-R)
Description: Leiter Scale is designed as nonverbal measure of intellectual function, memory and attention for Participants with communication disorders, hearing impairments, motor impairments, certain types of learning disabilities. Leiter-R was administered to participants after aging out of Bayley-III (at 42 months of age) and before Leiter-3 utilization (per protocol, due to discontinuation of Leiter-R). Leiter-R scale consists of 2 groups of subtests: Visualization-Reasoning Battery, Attention-Memory Battery. Subtests in Leiter-R were Figure Ground, Form Completion, Sequential Order, Repeated Patterns using that 'Brief Scale IQ' was scored for estimation of intellectual ability. Brief-IQ scores range is 30-170, where higher scores indicates higher intelligence. Score of 100 is expected mean standard score at each age interval. 95% children in each age group (based on normative sample) are expected to score within 2 SD of mean.
Time Frame: Participants 1 and 2: Week 156, Participant-3: Week 260, Participant-4: Week 156, Participant-5: Week 208
Population: Analysis was performed on FAS population. No summary analysis was done and participant wise data were reported at available specified timepoints (most recent visit). Here, "Overall number of participants analyzed" signifies participants who were evaluated for this outcome measure.
Measure: Number; unit: score on a scale
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 5
score on a scale
  Participant-1 Week 156: number analyzed (Participants) | 1
  Participant-1 Week 156 | 54
  Participant-2 Week 156: number analyzed (Participants) | 1
  Participant-2 Week 156 | 50
  Participant-3 Week 260: number analyzed (Participants) | 1
  Participant-3 Week 260 | 100
  Participant-4 Week 156: number analyzed (Participants) | 1
  Participant-4 Week 156 | 98
  Participant-5 Week 208: number analyzed (Participants) | 1
  Participant-5 Week 208 | 97

9. Primary Outcome: Nonverbal Intelligence Quotient (IQ) Score of Leiter International Performance Scale - 3rd Edition (Leiter-3)
Description: Leiter Scale: Designed as nonverbal measure of intellectual function, memory and attention for participants with communication disorders, hearing impairments, motor impairments, certain types of learning disabilities. Leiter-3 has 2 groups of subtests: cognitive battery and attention/memory battery. Nonverbal intelligence estimates global intellectual ability. The 4 cognitive battery subtests are: Figure Ground, Form Completion, Sequential Order, Classification-analogies along with 1 optional subset, Visual Patterns. Nonverbal IQ scores range is 30-170, which encompass 'severe delay' to 'extremely high/gifted', higher numbers indicates higher intelligence. Score of 100 is expected mean standard score at each age interval. 95% children in each age group (based on normative sample) are expected to score within 2 SD of mean.
Time Frame: Participant-1: Week 156, Participant-2: Week 312, Participant-3: Week 416
Population: Analysis was performed on FAS population. No summary analysis was done and participant wise data were reported at available specified timepoints (most recent visit). Here, "Overall number of participants analyzed" signifies number of participants who were evaluated for this outcome measure.
Measure: Number; unit: score on a scale
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 3
score on a scale
  Participant-1 Week 156: number analyzed (Participants) | 1
  Participant-1 Week 156 | 87
  Participant-2 Week 312: number analyzed (Participants) | 1
  Participant-2 Week 312 | 78
  Participant-3 Week 416: number analyzed (Participants) | 1
  Participant-3 Week 416 | 70

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: Adverse event (AE): any undesirable physical, psychological or behavioral effect experienced by participants during their participation in an investigational study, in conjunction with the use of the drug or biologic, whether or not product-related. Any untoward signs or symptoms experienced by the participant from the time of signing of the informed consent until completion of the study. Serious AE (SAE): any AE that resulted in any of the following outcomes: death, life-threatening experience, required hospitalization or prolonged inpatient hospitalization, persistent or significant disability/incapacity, congenital anomaly, and important medical events. TEAEs: AEs that developed, worsened, or became serious during the treatment-emergent period (defined as the period from the first study drug administration until last study assessment).
Time Frame: From Baseline up to 13.25 years
Population: Analysis was performed on FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 12
Participants
  TEAEs | 11
  TESAEs | 9

ADVERSE EVENTS:
Time Frame: From administration of first dose of study drug up to 13.25 years
Description: Reported AEs and deaths are TEAEs that developed, worsened, or became serious during the treatment period (from the first administration of study drug in the study to the last study assessment). Analysis was performed on FAS population.
Groups:
- Alglucosidase Alfa: Participants received alglucosidase alfa 20 mg/kg body weight as intravenous infusion every 2 weeks until 10 years of age or up to discontinuation from study treatment due to any reason.
Arm/Group | Alglucosidase Alfa
All-Cause Mortality (participants affected / at risk) | 3/12
Serious Adverse Events (participants affected / at risk) | 9/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alglucosidase Alfa (N=12)
Bacteraemia (Infections and infestations) | 1 (2)
Bronchitis (Infections and infestations) | 1 (1)
Catheter Site Infection (Infections and infestations) | 1 (1)
Device Related Sepsis (Infections and infestations) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Medical Device Site Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (18)
Pneumonia Aspiration (Infections and infestations) | 3 (4)
Pneumonia Bacterial (Infections and infestations) | 1 (1)
Pseudomonas Infection (Infections and infestations) | 1 (1)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Vascular Device Infection (Infections and infestations) | 5 (5)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Feeding Disorder (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemic Seizure (Nervous system disorders) | 2 (2)
Neurological Decompensation (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Bronchial Secretion Retention (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Velopharyngeal Incompetence (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1)
Glycogen Storage Disease Type Ii (Congenital, familial and genetic disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Oxygen Saturation Decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alglucosidase Alfa (N=12)
Ear Infection (Infections and infestations) | 2 (2)
Fungal Skin Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Oral Candidiasis (Infections and infestations) | 1 (2)
Otitis Media (Infections and infestations) | 6 (11)
Pharyngitis Streptococcal (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 6 (9)
Rash Pustular (Infections and infestations) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (13)
Urinary Tract Infection (Infections and infestations) | 2 (4)
Viral Pharyngitis (Infections and infestations) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (2)
Vulvovaginal Candidiasis (Infections and infestations) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1)
Allergy To Animal (Immune system disorders) | 1 (1)
Multiple Allergies (Immune system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Feeding Disorder (Metabolism and nutrition disorders) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Areflexia (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Focal Dyscognitive Seizures (Nervous system disorders) | 1 (1)
Hypotonia (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
White Matter Lesion (Nervous system disorders) | 1 (1)
Chalazion (Eye disorders) | 1 (1)
Eye Discharge (Eye disorders) | 2 (2)
Eye Swelling (Eye disorders) | 1 (1)
Eyelid Ptosis (Eye disorders) | 2 (2)
Papilloedema (Eye disorders) | 2 (2)
Visual Acuity Reduced (Eye disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
Deafness Neurosensory (Ear and labyrinth disorders) | 4 (4)
External Ear Disorder (Ear and labyrinth disorders) | 1 (1)
Middle Ear Effusion (Ear and labyrinth disorders) | 1 (1)
Right Ventricular Hypertrophy (Cardiac disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (17)
Flushing (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Bronchial Secretion Retention (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (28)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (16)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Velopharyngeal Incompetence (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (2)
Dental Caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (6)
Gingival Swelling (Gastrointestinal disorders) | 1 (1)
Mouth Ulceration (Gastrointestinal disorders) | 1 (1)
Post-Tussive Vomiting (Gastrointestinal disorders) | 1 (1)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1)
Swollen Tongue (Gastrointestinal disorders) | 1 (1)
Teething (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 7 (11)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (2)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 3 (5)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3)
Hair Growth Abnormal (Skin and subcutaneous tissue disorders) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (20)
Rash Papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Extremity Contracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint Contracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Catheter Site Rash (General disorders) | 1 (1)
Mass (General disorders) | 1 (1)
Pain (General disorders) | 4 (6)
Pyrexia (General disorders) | 9 (42)
Swelling (General disorders) | 1 (1)
Swelling Face (General disorders) | 1 (1)
Unevaluable Event (General disorders) | 1 (1)
Vascular Device Occlusion (General disorders) | 1 (1)
Audiogram Abnormal (Investigations) | 1 (1)
Bacterial Test Positive (Investigations) | 1 (1)
Blood Potassium Decreased (Investigations) | 1 (1)
Blood Urine Present (Investigations) | 1 (1)
Body Temperature Increased (Investigations) | 2 (2)
Clostridium Test Positive (Investigations) | 1 (2)
Electrocardiogram Qrs Complex Prolonged (Investigations) | 1 (1)
Electrocardiogram Qt Prolonged (Investigations) | 1 (1)
Electrocardiogram T Wave Inversion (Investigations) | 1 (1)
Fungal Test Positive (Investigations) | 1 (1)
Haematocrit Decreased (Investigations) | 1 (1)
Haemoglobin Decreased (Investigations) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 1 (5)
Pseudomonas Test Positive (Investigations) | 1 (1)
Tympanometry Abnormal (Investigations) | 1 (1)
Urine Output Decreased (Investigations) | 1 (1)
Anaesthetic Complication (Injury, poisoning and procedural complications) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1)
Stoma Site Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Device Malfunction (Product Issues) | 3 (4)

LIMITATIONS AND CAVEATS:
No summary analysis was done and participant wise data were reported at available specified timepoints. Reporting of participant numbers is per-endpoint and not consistent between assessments to maintain participant's privacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2014-12-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT00486889/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT00486889/SAP_001.pdf